CLINICAL TRIAL: NCT00151281
Title: Phase II Trial of Anti-Angiogenic Therapy With RT-PEPC in Patients With Relapsed Mantle Cell Lymphoma
Brief Title: Phase II Study of RT-PEPC in Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 047080073974
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: relapsed mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Prednisone; Cyclophosphamide; Etoposide; Procarbazine; Thalidomide; Rituximab

ARMS (1):
- Study Treatment Arm (Experimental)
  Interventions: Drug: PEPC; Drug: Thalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: PEPC — Induction phase (month 1-3)
  • PEPC daily (prednisone 20 mg/day, cyclophosphamide 50 mg/day, etoposide 50 mg/day, and procarbazine 50 mg/day) until expected drop in neutrophil count (ANC < 3000), unless due to disease. After ANC returns to above 2,000/ul, PEPC resumes at alternate day or fractionated weekly basis.
  Maintenance phase (month 4-12) • PEPC QOD or fractionated weekly basis.
  Post-Month 12 Maintenance phase (post-month 12 until disease progression)
  • PEPC QOD or fractionated weekly basis
  Other Names: Prednisone, Cyclophosphamide, Etoposide, Procarbazine
Drug: Thalidomide — Induction phase (month 1-3)
  • Daily thalidomide at 50 mg/day for the first 8 weeks, then dose escalated as tolerated to a maximum of 100 mg/day.
  Maintenance phase (month 4-12) • Daily low dose thalidomide (50-100 mg/d)
  Post-Month 12 Maintenance phase (post-month 12 until disease progression)
  • Daily low dose thalidomide (50-100mg/d)
Drug: Rituximab — Induction phase (month 1-3)
  • Rituximab weekly x 4 (375 mg/m2/week) starting at week 1.
  Maintenance phase (month 4-12) • Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months.
  Post-Month 12 Maintenance phase (post-month 12 until disease progression)
  • Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months

SUMMARY:
Primary Objective:

Evaluate the clinical activity of the RT-PEPC combination regimen (rituximab, thalidomide, and prednisone, etoposide, procarbazine, cyclophosphamide) in patients with relapsed mantle cell lymphoma. Specifically, response rate (RR) and time to disease progression (TTP) will be assessed.

Secondary Objectives:

1. Assess the toxicity profiles of RT-PEPC treatment in patients with relapsed mantle cell lymphoma.
2. Prospectively characterize the angiogenic profile of patients with mantle cell lymphoma during treatment with RT-PEPC. The dynamics of the angiogenic profile will be correlated with clinical response to RT-PEPC therapy.
3. Assess the quality of life of patients receiving RT-PEPC treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mantle cell Non-Hodgkin's Lymphoma with characteristic immunophenotypic profiles: CD5(+),CD23(-), CD19(+) or CD20(+), cyclin D1(+), and CD10(-)
* Patient has persistent / recurrent disease after standard chemotherapy
* Patient has not received either standard or investigational drugs within the last 3 weeks
* Available frozen tumor tissue obtained since completion of last prior therapy (rebiopsy if needed)
* Patient has measurable disease as defined by a tumor mass > 1.5 cm in one dimension
* Age > 18 years
* Absolute granulocyte count > 1000 cells/mm3
* Platelet count > 50,000 cells/mm3
* Creatinine < 2.0 x ULN
* Total bilirubin < 2.0 x ULN
* Patient has KPS > 50%
* Patient agrees to use birth control if of reproductive potential

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma
* Known HIV disease
* Known peripheral neuropathy > grade 2
* Patient is pregnant or nursing
* Patient has had major surgery within the last 3 weeks
* Patient is receiving other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2011-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Result] Ruan J, Martin P, Coleman M, Furman RR, Cheung K, Faye A, Elstrom R, Lachs M, Hajjar KA, Leonard JP. Durable responses with the metronomic rituximab and thalidomide plus prednisone, etoposide, procarbazine, and cyclophosphamide regimen in elderly patients with recurrent mantle cell lymphoma. Cancer. 2010 Jun 1;116(11):2655-64. doi: 10.1002/cncr.25055. PMID 20235190

RESULTS

PARTICIPANT FLOW:
Groups:
- RT-PEPC Drug Therapy: PEPC Induction phase PEPC daily (prednisone 20 mg/day, cyclophosphamide 50 mg/day, etoposide 50 mg/day, and procarbazine 50 mg/day) until expected drop in neutrophil count (ANC < 3000), unless due to disease. After ANC returns to above 2,000/ul, PEPC resumes at alternate day or fractionated weekly basis Maintenance phase PEPC QOD or fractionated weekly basis. Post-Month 12 Maintenance phase PEPC QOD or fractionated weekly basis Thalidomide Induction phase Daily thalidomide at 50 mg/day for the first 8 weeks, then dose escalated as tolerated to a maximum of 100 mg/day.
  Maintenance phase Daily low dose thalidomide (50-100 mg/d) Post-Month 12 Maintenance phase Daily low dose thalidomide (50-100mg/d) Rituximab Induction phase Rituximab weekly x 4 (375 mg/m2/week) starting at week 1. Maintenance phase Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months. Post-Month 12 Maintenance phase Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months
Period: Overall Study
Arm/Group | RT-PEPC Drug Therapy
Started | 25
Completed | 22
Not Completed | 3
Not completed — Not evaluable | 3

BASELINE CHARACTERISTICS:
Arm/Group | RT-PEPC Drug Therapy
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 68 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival and Progression Free Survival
Description: measured by overall Response Rate (ORR), which includes Complete response and partial response.
Time Frame: 38 months
Population: Twenty-five patients were enrolled, and 22 of those patients were assessable for response (3 patients were enrolled but received no therapy)
Measure: Number; unit: percentage of patients
Groups:
- Study Treatment Arm: Rituximab, Thalidomide, Prednisone, Etoposide, Procarbazine, Cyclophosphamide: Induction phase (month 1-3)
  * PEPC daily (prednisone 20 mg/day, cyclophosphamide 50 mg/day, etoposide 50 mg/day, and procarbazine 50 mg/day) until expected drop in neutrophil count (ANC < 3000), unless due to disease. After ANC returns to above 2,000/ul, PEPC resumes at alternate day or fractionated weekly basis.
  * Daily thalidomide at 50 mg/day for the first 8 weeks, then dose escalated as tolerated to a maximum of 100 mg/day.
  * Rituximab weekly x 4 (375 mg/m2/week) starting at week 1.
  Maintenance phase (month 4-12)
  * Daily low dose thalidomide (50-100 mg/d)
  * PEPC QOD or fractionated weekly basis.
  * Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months.
  Post-Month 12 Maintenance phase (post-month 12 until disease progression)
  * Daily low dose thalidomide (50-100mg/d)
  * PEPC QOD or fractionated weekly basis
  * Rituximab (375 mg/m2/week) weekly x 4 administered every 4 months
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 22
percentage of patients | 73

2. Secondary Outcome: Asses the Toxicity Profiles
Description: Toxicities were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0.
Time Frame: 38 months
Population: patients treated with study drug
Measure: Count of Participants; unit: Participants
Arm/Group | RT-PEPC Drug Therapy
Number analyzed (Participants) | 22
Participants
  Grade 3 or 4 neutropenia | 14
  Anemia | 1
  Thrombocytopenia | 4
  Fatigue | 22
  Constipation | 14
  Cough | 14
  Nausea | 13
  Neuropathy | 13
  Dyspnea | 11
  Rash | 10

3. Secondary Outcome: Dynamic Levels of Plasma VEGF
Description: Stromal angiogenesis was assessed using blood vascular and perivascular markers, including VEGFR-1, VEGFR-2, CD34, and a-SMA, as well as lymphatic vascular markers ofVEGFR-3, podoplanin, and Lyve-1.
Time Frame: 38 months
Population: subjects with evaluable VEGF level at baseline
Measure: Median (Full Range); unit: pg/mL
Arm/Group | RT-PEPC Drug Therapy
Number analyzed (Participants) | 20
pg/mL | 109.5 [7 to 319]

4. Secondary Outcome: The Quality of Life (QoL) of Patients Receiving RT-PEPC Treatment
Description: QoL assessments were obtained with version 3 of the Functional Assessment of Cancer Therapy-General (FACT-G) instrument. The FACT-G is comprised of four subscales: physical well-being (7-items, score range 0-28), social/family well-being (7-items, score range 0-28), emotional well-being (6-items, score range 0-24), and functional well-being (7-items, score range 0-28). Users of the FACT-G are able to generate an overall score and four subscale scores with ranges and distributions that are sample-specific. All questions in the FACT-G use a 5-point rating scale (0 = Not at all to 4 = Very much) A higher number indicates a better Quality of Life, and has a possible range of 0-108 points.
  ANOVA was used to compare the difference in the means of total score among the different time points (baseline, every 2M until 6M, and every 6M until PD). The mean of the total FACT-G scores at baseline and mean of total score at all timepoints (using ANOVA) are reported below.
Time Frame: baseline, every 2 months until Month 6, and every 6 months until disease progression
Measure: Mean (Full Range); unit: FACT-G score
Arm/Group | RT-PEPC Drug Therapy
Number analyzed (Participants) | 22
FACT-G score
  Mean FACT-G Score at baseline | 83.3 [64.5 to 102.1]
  Mean Total FACT-G Score between all time points | 89.4 [83.9 to 94.9]

ADVERSE EVENTS:
Arm/Group | Study Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=22)
pneumocystis carinii pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment Arm (N=22)
Neutropenia (Blood and lymphatic system disorders) | 20
Anemia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Pneumonia/ Upper Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 9
Fever (General disorders) | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Opportunistic infection (General disorders) | 2
Fatigue (General disorders) | 22
Constipation (Gastrointestinal disorders) | 14
Cough (General disorders) | 14
Nausea (General disorders) | 13
Neuropathy (Nervous system disorders) | 13
Dyspnea (General disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 10
Dizziness (General disorders) | 10
Abdominal pain (General disorders) | 8
Alopecia (Immune system disorders) | 8
Vomiting (General disorders) | 6
Deep Vein Thrombosis/ pulmonary embolism (Blood and lymphatic system disorders) | 2
Transient ischemic attack (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes